CLINICAL TRIAL: NCT06989073
Title: Effect of Muscle Energy Technique in Children With Post Traumatic Elbow Stiffness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zainab Sayed Farghaly Farghaly, Physiotherapist at bani suef specialized hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET in elbow stiffness
Record Dates: First submitted 2023-12-11; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Elbow Injuries
Keywords: Muscle energy technique
MeSH Terms: conditions — Elbow Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional treatment (Active Comparator): Hot Pack, Range of Motion,Stretching Exercises and Strengthing Exercises
  Interventions: Procedure: Convenional treatment
- Muscle Energy Technique (Experimental): Muscle Energy Technique is soft tissue or joint technique used in treatment of musculoskeletal dysfunctions
  Interventions: Procedure: Muscle Energy Technique

INTERVENTIONS:
Procedure: Muscle Energy Technique — METs are soft tissue or joint techniques that are employed in the treatment of musculoskeletal dysfunctions.
  Arms: Muscle Energy Technique
Procedure: Convenional treatment — Hot pack, Range of Motion Exercises, Stretching Exercises and Strengthening exercises.
  Arms: Conventional treatment

SUMMARY:
To investigate the effect of muscle energy technique on children with post traumatic elbow stiffness on pain level, functional disability and range of motion.

DETAILED DESCRIPTION:
Elbow fractures are the most common pediatric fracture and one of the most common fractures involving the upper extremity. Although both pediatric and adult patients may suffer this type of injury, the frequency and type of fracture, as well as the treatment of these injuries, are distinct in both populations. Due to the anatomic complexity of the elbow, multiple structures including the trochlea of the humerus, the olecranon, and the radial head, may all be involved.

Radial head and neck fractures occur most frequently in children aged 7 years to 12 years. The majority of proximal radius fractures are radial neck fractures (89%), and these fractures occur more frequently in younger patients compared to radial head fractures. A concomitant fracture occurs in up to 39% of radial head or neck fractures, and can easily be missed on the initial interpretation of the radiographs.

Children with a proximal radius fracture present with symptoms of pain and limited range of motion after a fall or other type of trauma. Patients generally refuse to move the affected elbow. In some cases, pain may be referred to the wrist. Physical examination shows swelling, and pain exacerbated by motion, particularly with attempted pronation and supination. There is tenderness on palpation of the proximal radius.

Neurovascular examination should be performed, specifically considering the posterior interosseous nerve. Attention should also be paid to soft-tissue swelling to assess the rare risk of forearm compartment syndrome.

Childhood fractures are common with a lifetime risk of 42%-64% in boys and 27%-40% in girls.

One-third of children will suffer at least one fracture before age seventeen, and upper limb fractures account for 72.1% of these. Elbow fractures are common in pediatric populations. Hussain reported that 28.4% of all pediatric fractures were elbow fractures, which were the most common type of fractures.

The most common trauma mechanism for radial head and neck fractures is valgus loading with the elbow in extension, such as a fall on an outstretched hand. The force through the lateral capitulum compresses the radial head, causing it to break at the weakest point, which is often the radial neck at the metaphysis. A second injury mechanism is a radial head dislocation, which is most commonly seen in radial head fractures.

Elbow fracture mechanisms are classified into six categories as follows: tumble tumbled on the outstretched elbow at ground level; fall, fall on the outstretched elbow from above ground level; lateral bend, bent the elbow during sports or accidents; direct hit, smashed by an object or the elbow got caught in the door; throw, injured after throwing a ball or other object, and unknown. The etiologies were categorized by the activity or location of the injuries (e.g. tumble while playing football/skateboarding, fall from chair/bed, or lateral bend during Judo). There could be functional losses seen with even less severe loss of range of motion (ROM) at the elbow.

A stiff elbow has been defined as one with a loss of extension of greater than 30° and flexion of less than 120°. Restriction of joint mobility is a common complication that is seen post-elbow fracture. This could be due to immobilization, pain, muscle guarding, etc. All these may lead to reduced joint function and may restrict the patient's ability to perform functional tasks, thereby affecting his activities of daily living.

The muscle energy technique is a form of manual therapy widely used in Osteopathy, which uses a muscle's own energy in the form of gentle isometric contractions to relax the muscles via autogenic or reciprocal inhibition and lengthen the muscle.

As compared to static stretching which is a passive technique in which the therapist does all the work, MET is an active technique in which the patient is also an active participant. MET is based on the concepts of Autogenic Inhibition and Reciprocal Inhibition. If a sub-maximal contraction of the muscle is followed by stretching of the same muscle it is known as Autogenic Inhibition MET, and if a submaximal contraction of a muscle is followed by stretching of the opposite muscle then this is known as Reciprocal Inhibition MET MET involves the subject voluntarily contracting the muscle in a precisely controlled direction against the therapist's counterforce. Its therapeutic effects are to reduce pain, reduce muscle tone, stretch tightened muscles, strengthen weak muscles, improve local circulation, and mobilize joint restriction.

ELIGIBILITY:
Inclusion Criteria:

* Children from both gender.
* Age ranges from 6-12 years.
* Patients with post-traumatic elbow stiffness after distal end extra-articular humerus fractures.
* Patients with proximal radius ulna fractures.
* Minimum immobilization period of 4 weeks.
* Referred from orthopedist.
* Patient with soft end feel.

Exclusion Criteria:

* Any ligament injury
* Patients with Diabetes
* Patients with Rheumatoid Arthritis.
* Patients with Pathological fractures
* Revision surgeries
* Neuro-vascular disorders.
* Patient with bony end feel.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Investigate the effect of muscle energy technique on children with elbow stiffness | 4 weeks
  Measure range of motion with goniometer pro application
Investigate the effect of muscle energy technique on children with elbow stiffness | 4 weeks
  Measure Pain with Faces Pain Scale_Revised

SECONDARY OUTCOMES:
Investigate the effect of muscle energy technique on children with elbow stiffness | 4 weeks
  Measure Quality Of Life with Pediatric Quality Of Life Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Maher Alqabalawy, Prof. doctor, Study Chair — Cairo University; Sahar Abdallah, Professor, Study Director — Cairo University
Locations (1):
- Faculty of physical therapy, Cairo university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behdad A, Behdad S, Hosseinpour M. Pediatric elbow fractures in a major trauma center in iran. Arch Trauma Res. 2013 Winter;1(4):172-5. doi: 10.5812/atr.8098. Epub 2013 Feb 1. PMID 24396773